CLINICAL TRIAL: NCT04923997
Title: The HealthScore Health Coaching Program
Acronym: HealthScore
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LCCC 1948
Record Dates: First submitted 2021-06-07; First posted 2021-06-11 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Cancer; Survivorship; Quality of Life; Health Behavior
Keywords: Health Coaching; Wellness; Integrative
MeSH Terms: conditions — Neoplasms; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health Coaching (Experimental): All participants will be in the health coaching group. Participants on study will receive a health coach for 6 months.
  Interventions: Behavioral: Health Coaching

INTERVENTIONS:
Behavioral: Health Coaching — 6 months of integrative health coaching, goal setting, survey administration and physical assessments.

SUMMARY:
Purpose: The HealthScore Health Coaching Program aims to deliver 6-months of 1:1 home-based health coaching to cancer patients receiving treatment and survivors of any diagnosis at UNC Cancer Hospital. This study hopes to preserve physical function, address unmet physical, nutritional, psychological, social and other needs.

Procedures: This will be done through individualized health coaching, weekly symptom survey administration, monthly supportive care questionnaires, and physical assessments at baseline, 3 months and 6 months.

Participants: All cancer patients with appointments at UNC Cancer Hospitals.

DETAILED DESCRIPTION:
Evaluation and monitoring are used sporadically in routine cancer care, and cancer coaching programs are rare. The potential for these approaches to improve quality of life and clinical outcomes in cancer patients is significant. The HealthScore Health Coaching Program is designed as a way to routinely combine evaluation, monitoring and coaching within a single framework as a six-month intervention for cancer patients or survivors. The primary rationale for the Program is that improvements in physical function, unmet needs identification, and self-efficacy are likely to lead to better patient-centered and overall outcomes for patients and survivors. A secondary rationale is that the framework of the Program and data obtained as part of the Program will facilitate additional quality improvement and research activities to refine the application of evaluation, monitoring and coaching techniques in cancer care. As reimbursement and care delivery in oncology transition to a focus on value and population-based management, the HealthScore Health Coaching Program may provide a model for application to cancer care within and outside UNC. The primary purpose of this study is to provide 6-months of 1:1 home-based health coaching for cancer patients and survivors will improve physical function and address unmet physical, nutritional, psychological, social and other needs which will increase patient and survivor self-efficacy for medical engagement, reduce morbidity, health care utilization, and encourage health lifestyle behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have an appointment at a cancer center, including if they are an inpatient, if they are seen by a clinical service providing care to patients with cancer or sickle cell disease, and if they are > age 15. They can be receiving active treatment or in survivorship, with no restrictions based on time since the conclusion of active treatment. No exclusions will be made based on gender, ethnicity or race.
* Patient must be willing and able to participate in a 6-month intervention.
* Patients must be willing and able to provide patient-reported survey responses electronically or by telephone.
* Patients must have the ability to use a wearable sensor and view wearable sensor data at home.
* Patients must have a working email address and have the ability to check and respond to email.
* Participation in a research study is allowable by the patient's insurance provider

Exclusion Criteria:

* Patients who do not read and speak English, as program software has not been translated into other languages at this time.
* The patient has concurrent medical or psychiatric conditions that may preclude participation (i.e. moderate to severe dementia, uncontrolled schizophrenia, or other conditions that would render them unable to provide informed consent or complete questionnaires).

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2025-05-11 (Actual); Study Completion 2025-05-11 (Actual)

PRIMARY OUTCOMES:
Percent Completion | 5 years
  To provide health coaching services for cancer patients and survivors at UNC through the HealthScore Program, measured by calculating numbers of participants enrolled and completing the six-month HealthScore health coaching intervention each year.

SECONDARY OUTCOMES:
Change in Physical Function | 6 months
  Change in PROMIS (Patient Reported Outcomes Measurement Information System) Physical Function 8b on a scale of 0-60.5. Higher scores indicate better physical function.
Completed coaching phone calls | 6 months
  Percentage of possible coaching phone calls completed
Survey Completion | 6 months
  Percentage of possible patient-reported surveys completed
Wearable Sensor data | 6 months
  Percentage of possible days using the wearable sensor with evaluable data
Unmet Needs | 6 months
  Number of unmet needs addressed while participating in health coaching
Change in participant self-efficacy using the Lorgis Self-Efficacy Scale | 6 months
  Magnitude of change in self-efficacy during program participation using the Lorgis Self-efficacy scale. The score is the mean of six items, scored 0-10. Higher scores are better.

CONTACTS AND LOCATIONS:
Overall Officials: William A Wood, MD, MPH, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Khairat S, Kent EE, Geracitano J, Mendis K, Zhou Z, Bailey C, Wood WA. Efficacy of Telehealth-Based Coaching to Improve Physical Activity and Overall Experience for Cancer Survivors: Secondary, Mixed Methods Analysis of a Randomized Controlled Trial. JMIR Cancer. 2026 Jan 15;12:e78968. doi: 10.2196/78968. PMID 41538790
- [Derived] Wood WA, Bailey C, Castrogivanni B, Mehedint D, Bryant AL, Lavin K, Tan X, Richardson J, Qian Y, Tan KR, Kent EE. Piloting HealthScore: Feasibility and acceptability of a clinically integrated health coaching program for people living with cancer. Cancer Med. 2023 Apr;12(7):8804-8814. doi: 10.1002/cam4.5625. Epub 2023 Jan 16. PMID 36647557